CLINICAL TRIAL: NCT00442130
Title: Reduced Intensity Stem Cell Transplantation for Advanced Chronic Lymphocytic Leukemia Followed by Vaccination With Lethally Irradiated Autologous Tumor Cells Admixed With Granulocyte Macrophage-colony Stimulating Factor Secreting K562 Cells
Brief Title: Reduced Intensity Stem Cell Transplantation for Chronic Lymphocytic Leukemia Followed by Vaccination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Catherine Wu, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-196
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: GM-CSF; GM-K562; vaccine
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GM-K562 Vaccine (Experimental): Biological/Vaccine: GM-K562 vaccine The vaccine will be administered over 1 cycle of 7 weeks, that begins 1 month after stem cell transplant. The vaccine will be given 6 times over 2 months -- once a week for three weeks then every other week for 3 vaccines.
  Procedure/Surgery: stem cell transplantation Participants will be admitted to the hospital for approximately 8 days to receive chemotherapy and stem cell transplantation
  Interventions: Biological: GM-K562 vaccine; Procedure: stem cell transplantation

INTERVENTIONS:
Biological: GM-K562 vaccine — The vaccine will be administered over 1 cycle of 7 weeks, that begins 1 month after stem cell transplant. The vaccine will be given 6 times over 2 months -- once a week for three weeks then every other week for 3 vaccines.
Procedure: stem cell transplantation — Participants will be admitted to the hospital for approximately 8 days to receive chemotherapy and stem cell transplantation

SUMMARY:
The purpose of this research study is to assess the safety and immune activity of a vaccine made from the participant's own cancer cells, when administered after a reduced intensity transplant. In recent years, researchers at Dana-Farber Cancer Institute have discovered that vaccines made from a patients's own cancer cells, that have been engineered in the laboratory to produce a protein called GM-CSF, can be effective in stimulating a powerful immune response specific to that cancer.

DETAILED DESCRIPTION:
* This study can be divided into four phases: 1) Screening; 2) Reduced intensity transplant phase; 3) Vaccinations (cycle 1 and cycle 2:each cycle lasts 7 weeks) and 4) Vaccine completion.
* Screening Phase: After signing the consent form, participants will be asked to undergo some screening tests and procedures to find out if they are eligible to participate in the study. These tests and procedures are likely to be part of regular cancer care and may be done even if the patient does not take part in the research study. It is important to note that if insufficient numbers of the participant's leukemia cells to generate vaccine were collected on the CLL collection and banking study (DF/HCC study 06-200), then they will not be eligible to participate in this study.
* Allogeneic reduced intensity stem cell transplant phase: The transplant phase of the study will begin when the participant is admitted to the hospital to receive chemotherapy and stem cell transplant. The minimum duration of hospitalization for the procedure is approximately 8 days. Undergoing transplant involves the following procedures and treatments: Central intravenous catheter; chemotherapy; medications to prevent graft versus host disease (GVHD); medication to prevent infections; physical exams; blood tests and bone marrow biopsy and aspirate.
* Vaccination Phase: Vaccinations will be given in two cycles, of seven weeks each, that are identical with the exception of when they are administered. Cycle 1 vaccination will begin approximately one month after the stem cells have been infused, provided there is no significant evidence of GVHD. Cycle 2 vaccination will be being approximately one month after discontinuing tacrolimus, provided there is no evidence of severe acute or chronic GVHD. The vaccine will be given 6 times over a period of two months. The participant will receive vaccination shots once weekly for 3 vaccines and then every other week for 3 vaccines.
* Skin biopsies will be done after the first and after the fifth vaccinations. Current status of the participants CLL will be assessed to determine how the disease has responded to transplant and vaccination. These tests include analysis of bone marrow and blood tests.
* Vaccine completion phase: After one cycle of vaccination is completed, the participant will return to the outpatient clinic monthly for check-ups for 6 visits, to monitor the effects of the vaccine.
* Since this trial involves the use of genetically modified cells, it is recommended that participants on this trial undergo annual checkups for at least 20 years, in order to monitor for long term effects of the vaccination treatment.

ELIGIBILITY:
Inclusion Criteria:

* Advanced CLL, defined as no response or progressive disease during standard nucleoside analogue based regimen; or, evidence of progressive disease within 24 months of completion of nucleoside analogue regimen; or, intolerance to fludarabine; or, failure to achieve complete remission following salvage regimen.
* no sites of adenopathy > 5cm
* (8/8) HLA matched related or unrelated donor available.
* Must have prior banked tumor, collected by peripheral blood draw, leukapheresis, bone marrow biopsy or by lymph node dissection, per DF/HCC protocol 06-200
* ECOG performance status 0-2

Exclusion Criteria:

* Serum creatinine greater than or equal to 2.0mg/dl
* ALT or AST greater than or equal to 3x ULN
* Total bilirubin greater than or equal to 2.0mg/dl (except for patients with Gilbert's syndrome)
* Cardiac ejection fraction greater than or equal to 30%
* HIV infection
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-02; Primary Completion 2014-02 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
To assess the safety and toxicity of vaccination with lethally irradiated autologous CLL cells admixed with GM-562 cells following reduced intensity allogeneic stem cell transplant for CLL patients with advanced disease. | 2 years

SECONDARY OUTCOMES:
To characterize the biologic activity in response to vaccination with lethally irradiated autologous CLL cells admixed with GM-562 cells, following reduced intensity allogeneic stem cell transplant | 2 years
to estimate duration of disease response, disease free and overall survival. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J. Wu, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Burkhardt UE, Hainz U, Stevenson K, Goldstein NR, Pasek M, Naito M, Wu D, Ho VT, Alonso A, Hammond NN, Wong J, Sievers QL, Brusic A, McDonough SM, Zeng W, Perrin A, Brown JR, Canning CM, Koreth J, Cutler C, Armand P, Neuberg D, Lee JS, Antin JH, Mulligan RC, Sasada T, Ritz J, Soiffer RJ, Dranoff G, Alyea EP, Wu CJ. Autologous CLL cell vaccination early after transplant induces leukemia-specific T cells. J Clin Invest. 2013 Sep;123(9):3756-65. doi: 10.1172/JCI69098. Epub 2013 Aug 5. PMID 23912587